CLINICAL TRIAL: NCT00714129
Title: De Novo Lipogenesis, Lipid and Carbohydrate Metabolism in Non-alcoholic Fatty Liver Disease
Acronym: LINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Touro University (Other); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DK078133-01 (NIH); NIH R01DK078133-01A1; ADA 1-08-CR-56
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Non-alcoholic Fatty Liver Disease; Diabetes
Keywords: Steatosis; Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus; Fatty Liver | interventions — Diet Therapy; Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Weight loss diet - normal diet
  Interventions: Other: Dietary intervention (calorie restricted diet)
- 2 (Experimental): Weight loss diet - low in simple sugars (specifically fructose)
  Interventions: Other: Dietary intervention (calorie restricted diet)

INTERVENTIONS:
Other: Dietary intervention (calorie restricted diet) — Participants in Aim 2 will receive a calorie restricted diet. This group will receive all their food for approximately 8 weeks which is the similar composition of their current diet.
  Arms: 1
Other: Dietary intervention (calorie restricted diet) — Participants in Aim 2 will receive a calorie restricted diet. This group will receive all their food for approximately 8 weeks which is lower in simple sugars, specifically fructose.
  Arms: 2

SUMMARY:
The worldwide epidemic of obesity is paralleled with increased cases of non-alcoholic liver disease (liver fat accumulation) and diabetes. Fat belongs in the adipose tissue, and if excess fat accumulates in the liver or muscle, these tissues cannot use sugar efficiently. It has been discovered that when large quantities of fructose (a sugar present in soft drinks) are consumed, the conversion of carbohydrate (CHO) to fat in the liver increases.

We hypothesize that: 1) subjects with fatty liver have a higher CHO uptake and conversion to fat in their liver when compared to matched control subjects with normal liver fat content; and that: 2) when subjects with fatty liver are fed a diet limiting fructose and simple sugars will decrease their liver CHO fat content. This reduction in liver fat will normalize the way the liver responds to sugar and insulin, reversing the pre-diabetic state.

The measurement of these parameters will be done using state-of-the-art techniques such as safe non-radioactive isotope tracers and non-invasive magnetic resonance spectroscopy.

For more information, please call 415-206-5532 for a phone screening

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common liver ailment in developed countries. Fatty liver - steatosis - affects up to one third of the population. Its prevalence is rising and seems to parallel the global increase in obesity and type-2 diabetes. The etiology of NAFLD in humans is not well understood. We propose that the hepatic conversion of carbohydrates (CHO) to lipids (de novo lipogenesis, DNL) is a key factor in the accumulation of excess liver fat and the accompanying dyslipidemia and hepatic insulin resistance; and that suppressing DNL by diet will reduce liver fat and improve both lipid and carbohydrate metabolism in patients with steatosis. These hypotheses are based on studies in which we and others have established that fractional hepatic DNL can vary dramatically depending on the diet and/or health status of a subject; and, in particular, that dietary fructose is a potent lipogenic stimulus. In this proposal we will perform CRC-based studies to compare the rates of DNL and very low density lipoprotein (VLDL) kinetics in steatotic and matched non-steatotic controls and evaluate their relationship to lipid profiles and hepatic and whole-body insulin resistance and overall carbohydrate metabolism (Aim1). The steatotic individuals whose habitual intake of fructose and other simple sugars exceeds 15% of total energy intake will then be randomized to consume one of two low-fat diets that differ only in CHO type to determine whether diet-induced changes in DNL affect liver fat flux and content and hepatic, whole-body insulin sensitivity, and overall carbohydrate metabolism (Aim 2). We hypothesize that a diet that is rich in complex CHO will achieve greater decreases in DNL and liver fat than one that contains typical amounts of simple CHO, including fructose. This dietary intervention study includes a 6-week 25% energy restriction outpatient phase to promote moderate weight loss and improve insulin sensitivity, followed by a two weeks weight maintenance with the last 4 days as an inpatient stay during which all of the studies performed at baseline (Aim 1) will be repeated. State-of-the-art stable isotope techniques will be used to assess hepatic DNL, apoB100 turnover, VLDL-triglyceride (TG) fluxes, and lipolysis under fasting and fed conditions. Hepatic and extra-hepatic insulin sensitivity will be measured using hyperinsulinemic-euglycemic clamps and stable isotope studies of endogenous glucose production and glycogen flux. Liver and muscle fat will be measured by proton magnetic resonance spectroscopy (MRS), visceral fat by magnetic resonance imaging (MRI), and whole-body composition by dual-energy X-ray absorptiometry (DEXA). These studies will allow us to evaluate the importance of DNL as a mechanism modulating liver fat content and flux, and the significance of CHO quality in dietary guidance for steatotic patients.

ELIGIBILITY:
Inclusion Criteria:

* In the steatotic subjects, steatosis will be diagnosed by MRS or liver biopsy in which >33% of the hepatocytes will contain fat. Non-steatotic controls will not have biopsies since they are not medically warranted; thus, to ensure they do not have steatosis they will undergo MRS during screening and have a total lipid: unsuppressed water < 0.05.

Exclusion Criteria:

* Habitual consumption of alcohol > 20 g/day for men and 10 g/day for women
* Confirmed HIV-1 infection, Hgb <13 g/dL for males and <12 g/dL for females
* Abnormal hepatitis B or C serology
* Diabetes or current use of any antidiabetic or hypolipidemic agents
* Presence of metal-containing substances in the body (e.g. a fragment in the eye, aneurysm clips, ear implants, spinal nerve stimulators or a pacemaker)
* Weight over 350 pounds or severe claustrophobia, which would preclude the MR studies
* Any condition that would preclude adherence to the protocol or the ability to provide informed consent
* Change in body weight >5% within the preceding 6 months (by self-report)
* Known intolerance, allergy or hypersensitivity to fructose
* Pregnancy or lactation (for women); OR
* Any other condition that, in the opinion of the investigators, would put the subject at risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2007-09; Primary Completion 2012-10-12 (Actual); Study Completion 2012-10-12 (Actual)

PRIMARY OUTCOMES:
Stable isotopic and magnetic resonance measures to determine the changes in lipid and carbohydrate metabolism after dietary intervention | approximately 8 weeks

SECONDARY OUTCOMES:
DEXA, insulin sensitivity and energy expenditure changes due to dietary intervention | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Schwarz, PhD, Principal Investigator — Touro University and UCSF
Locations (1):
- Touro University, Vallejo, California, United States